CLINICAL TRIAL: NCT07017569
Title: Design and Development of an Interactive Mobile Health (mHealth) App to Provide Momentary and Periodic Intervention for High Anxiety and Depression
Brief Title: An Interactive Mobile Health (mHealth) App as Intervention for High Anxiety and Depression in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2020-0162DCR
Record Dates: First submitted 2025-05-16; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Depression - Major Depressive Disorder; Stress
Keywords: Machine Learning; Mobile Health; Psychological Stress; Wearable Devices; College Students
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a 3:1 ratio into intervention and control groups respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital intervention (Experimental): This group will receive the mHELP mobile and watch application with full functionality which provides weekly self-assessment and self-reported events PLUS self-management functionality. The self- management functionality includes additional on-demand features.
  Interventions: Behavioral: Mobile health application
- Non intervention (No Intervention): This group will receive an Apple Watch and an iPhone mobile application to 1) complete weekly assessments of their mental health using PSS-10, GAD-7, and PHQ-9, and 2) to self-report high-anxiety or high- stress events. The mobile or watch applications will not have any other functionality. This version of the app will also include information about mental health resources provided to them on TAMU campus.

INTERVENTIONS:
Behavioral: Mobile health application — This group will receive the mHELP mobile and watch application with full functionality which provides weekly self-assessment and self-reported events PLUS self-management functionality. The self- management functionality includes additional on-demand features (see the attached list of features). These include
  * a breath functionality that provides a times breathing exercise similar to the one provided by the Apple iWatch; users can see changes in their heart rate during the breathing exercise and will see a summary of heart rate changes
  * a calendar features that allows students to upload their class schedule and see different activities such as self-assessments
  * a journaling feature that allows participants to write a journal
  * a task list to take note of major tasks and add them to calendar
  * a set of relaxation media including videos and audios that participants can use on demand
  Arms: Digital intervention

SUMMARY:
The goal of this clinical trial is to learn if a mobile health app called mHELP can help college students manage anxiety, stress, and depression.

The main questions it aims to answer are:

* Does using the mHELP app reduce anxiety, stress, and depression symptoms both over time and in real-time?
* Does the app help students engage with mental health services and self-management tools?

Researchers will compare students who use the full version of the mHELP app to those who use a control version with limited features.

Participants will:

* Use an Apple Watch and iPhone app for 10 weeks
* Receive reminders to complete weekly mental health questionnaires
* Tap a button to report high-stress moments or respond to automatic alerts from the app
* Intervention group will use app features like breathing exercises, journaling, and educational videos
* Intervention group will receive 2 free telehealth counseling sessions

DETAILED DESCRIPTION:
There will be two groups of participants:

1. Control (n=50): This group will receive an Apple Watch and an iPhone mobile application to 1) complete weekly assessments of their mental health using PSS-10, GAD-7, and PHQ-9, and 2) to self-report high-anxiety or high- stress events. The mobile or watch applications will not have any other functionality. This version of the app will also include information about mental health resources provided to them on TAMU campus.
2. Intervention (n=150): This group will receive the mHELP mobile and watch application with full functionality which provides weekly self-assessment and self-reported events PLUS self-management functionality. The self- management functionality includes additional on-demand features (see the attached list of features). These include

   * a breath functionality that provides a times breathing exercise similar to the one provided by the Apple iWatch; users can see changes in their heart rate during the breathing exercise and will see a summary of heart rate changes
   * a calendar features that allows students to upload their class schedule and see different activities such as self-assessments
   * a journaling feature that allows participants to write a journal
   * a task list to take note of major tasks and add them to calendar
   * a set of relaxation media including videos and audios that participants can use on demand No data will be collected on these activities except for overall usage time to assess engagement.

At the beginning of the study, participants in the intervention group are required to schedule and attend an introductory session with TAMU Telehealth Clinic. This service uses a video communication tool called MEND. mHELP provides a link to MEND registration but does collect any data about the telehealth sessions or any other information related to these visits. After their introductory session, participants are also required to schedule and attend a full session using MEND. If the participant wishes to continue using the telehealth services, they are allowed to do so, but it is not required. The telehealth clinic is staffed by qualified therapists from Texas A&M Telehealth Clinic.

The intervention group will also follow a case-control design for digital coaching/education: The first 5 weeks, participants will have access to educational content on demand. The second 5 weeks, participants will receive daily reminders to complete educational modules (e.g., short videos, posters, articles).

Each week will cover a different topic related to mental health:

Week 1 - Anxiety Week 2 - Sleep Week 3 - Depression Week 4 - Stress Week 5 - Grief/Relationships The purpose of the videos, posters, and articles provided is to help participants identify, recognize symptoms, and cope with each topic. The information was extracted from the TAMU Counseling and Psychological Services (CAPS) website.

Participants will be provided with consent forms prior to the start of any aspect of the study explaining the risks, benefits, time commitment. The study will start in late September and last until the last day of classes (10 weeks). Demographic information will be collected at the start of the study, including health, fitness status and lifestyle questionnaires. Students will be provided with a smartwatch and smartphone app, designed for convenient and momentary collection of self-reported events, and will be asked to wear the smartwatch continuously for the duration of the study. Participants will receive virtual instructions and practice on momentary assessments to enable self-reporting of anxiety and depression triggers. Participants will be instructed to tap anywhere on the smartwatch screen whenever they feel or perceive high anxiety and depression levels. Also, participants will receive notifications of stress moments detected by machine learning algorithms and respond to the notifications regarding whether the detection was correct or not. In addition, the investigators will obtain daily sleep logs via a smartphone app entry. At the start, middle, and end of the week, participants will be instructed to fill short online questionnaires on anxiety (using the Generalized Anxiety Disorder 7-item [GAD-7]), depression (using the Patient Health Questionnaire [PHQ-9], stress (using the 10-item Perceived Stress Scale [PSS-10]) and physical activity. Finally, participants will fill out a survey on intervention effectiveness pre-, mid-, and post-study. Periodic text reminders will be sent to participants to log the associated study measures via the smartphone app and will also add descriptions related to digital health coaching. A short exit interview will be conducted to collect information on students' experience with the app.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be 18 years or older.
* Participants should have an iPhone with at least iOS14
* Participants recently sought out resources to help with mental health problems they have experienced.
* Participants must score above a 7 on the GAD-7, to indicate probably Generalized Anxiety Disorder and at least moderate anxiety symptoms.
* Participants should be able to communicate in English.

Exclusion Criteria:

* Participants should not have severe anxiety/panic attacks, a history of suicidal attempt, current suicidal ideation, or current self-harm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Machine Learning detected Stress Moments | From enrollment through completion of the study, an average of 12 weeks
  The primary dependent variable, "Moments of Stress" (MS), is a conceptual real-time measure derived from a combination of physiological heart rate (beats per minute - bpm) measurements and subjective self-reports, both collected through the mHELP application on the Apple Watch. Participants were prompted by the app after periods of elevated heart rate, identified using an integrated machine learning algorithm, to provide momentary self-assessments of stress using a single-item scale (e.g., "Are you feeling stressed right now?"), enabling an acute, context-sensitive capture of perceived stress.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Weekly through study completion, an average of 12 weeks
  A subjective measure of stress and psychological functioning, the PSS, was collected as a secondary outcome measure. Once a week, the mHELP app would prompt the students to take these psychological surveys. The PSS has a minimum score of 0 and a maximum score of 40, with a higher score indicating higher general perceived stress.
Generalized Anxiety Disorder 7-item Scale (GAD-7) | Weekly through study completion, an average of 12 weeks
  A subjective measure of anxiety and psychological functioning, the GAD-7, was collected as a secondary outcome measure. Once a week, the mHELP app would prompt the students to take these psychological surveys. The GAD-7 has a minimum score of 0 and a maximum score of 21, with a higher score indicating higher symptoms of anxiety.
Patient Health Questionnaire - 8 (PHQ-8) | Weekly through study completion, an average of 12 weeks
  A subjective measure of depression and psychological functioning, the PHQ-8, was collected as a secondary outcome measure. Once a week, the mHELP app would prompt the students to take these psychological surveys. The PHQ-8 has a minimum score of 0 and a maximum score of 24, with a higher score indicating higher symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Farzan Sasangohar, Ph.D. Industrial Engineering, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared in this study as we plan to keep the personalized data private within the research personnel on the approved protocol. Rather, aggregate data will be published via journal article.